CLINICAL TRIAL: NCT02101944
Title: Pilot Trial Evaluating Viral Protein Production From the Combination of Reolysin and Carfilzomib in Multiple Myeloma
Brief Title: Wild-Type Reovirus in Combination With Carfilzomib and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00643; NCI-2014-00643 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-14031; 14031; NCI-9603; 2014C0091; 9603 (Other: Emory University Hospital/Winship Cancer Institute); 9603 (Other: CTEP); P30CA016058 (NIH); U01CA076576 (NIH); UM1CA186691 (NIH); UM1CA186712 (NIH)
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Anemia; Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Anemia; Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dexamethasone, carfilzomib, Reolysin) (Experimental): Patients receive dexamethasone intravenously (IV), carfilzomib IV over 30 minutes, and Reolysin IV over 60 minutes on days 1, 2, 8, 9, 15, and 16. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Biological: Pelareorep

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Carfilnat; CFZ; Kyprolis; PR-171
Drug: Dexamethasone — Given IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pelareorep — Given IV
  Other Names: PO BB0209; PO-BB0209; Reolysin; Reovirus Serotype 3; Wild-type Reovirus

SUMMARY:
This phase I trial studies the side effects and best dose of wild-type reovirus when combined with carfilzomib and dexamethasone in treating patients with multiple myeloma that has come back following treatment (relapsed) or does not respond to treatment (refractory). Chemotherapy drugs, such as dexamethasone and carfilzomib, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. A virus called wild-type reovirus may be able to kill cancer cells without damaging normal cells and seems to work best when given with chemotherapy. Giving wild-type reovirus with chemotherapy may be a more effective treatment than chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine safety and tolerability, and define the maximum tolerated dose of pelareorep (Reolysin), carfilzomib and dexamethasone in patients with relapsed multiple myeloma.

II. Obtain evidence of reovirus entry into myeloma cells via localization of reoviral ribonucleic acid (RNA) in multiple myeloma (MM) cells (in situ hybridization [ISH]), and active viral proliferation/replication via localization of reoviral capsid protein (immunohistochemistry [IHC]) in MM cells in cycle 1 day 9 bone marrow biopsies in all patients enrolled in dose escalation cohorts.

SECONDARY OBJECTIVES:

I. Obtain preliminary data on response as determined by International Myeloma Working Group criteria after protocol therapy.

II. Obtain overall and progression free survival data for all treated patients. III. Assess cytokine arrays of peripheral blood obtained on days 1, 2, 9, 15 and once during days 22-28 of cycle 1, and day 1 of cycle 2 and each successive cycle to obtain exploratory data regarding inflammatory cytokine concentrations and their correlation with response.

IV. Investigate pretreatment cycle 1 days 1 and 9 bone marrow aspirate interferon (IFN)-beta in MM cells as a potential marker of Reolysin resistance.

V. Measure the induction of endoplasmic reticulum (ER) stress and autophagy markers to explore their respective roles in MM cell death following combination Reolysin and carfilzomib in patients treated in all dose escalation cohorts.

VI. Evaluate pretreatment cycle 1 days 1 and 9 peripheral blood to explore the antiviral humoral response by measuring the production of neutralizing reoviral antibody (NARA) using a functional killing assay.

VII. Obtain cycle 1 day 1 pretreatment and 1 and 4 hours after treatment, and pretreatment cycle 1 days 2 and 9 peripheral blood, and pretreatment cycle 1 days 1 and 9 bone marrow aspirate samples to investigate the role of carfilzomib in modulating the antiviral immune mediated response.

OUTLINE: This is a dose escalation study of Reolysin.

Patients receive dexamethasone intravenously (IV), carfilzomib IV over 30 minutes, and Reolysin IV over 60 minutes on days 1, 2, 8, 9, 15, and 16. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have relapsed or refractory myeloma that fits or did fit International Myeloma Working Group (IMWG) diagnostic criteria for symptomatic myeloma (although new or worsening end organ damage is not required to be eligible) as defined below:

  * Presence of clonal bone marrow plasma cells
  * Evidence of any end organ damage criteria listed below (at any time) attributed to the patient's myeloma:

    * Hypercalcemia: serum calcium > 11.5 mg/dL or
    * Renal insufficiency: serum creatinine > 2 mg/dL
    * Anemia > 2 g/dL below the lower limit of normal or a hemoglobin value < 10 g/dL
    * Bone lesions: lytic lesions, severe osteopenia or pathologic fractures
* In the safety expansion 10 patient group but not during dose escalation, patients must have measurable disease defined as any of the following:

  * Serum monoclonal protein >= 500 mg/dL by protein electrophoresis
  * > 200 mg of monoclonal protein in the urine on screening 24-hour electrophoresis
  * Serum immunoglobulin free light chain >= 100 mg/L AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Patients must have been previously treated with an immunomodulatory drug (IMiD) and proteasome inhibitor, must be refractory to carfilzomib defined as progression on or within 2 months of a carfilzomib-containing therapy, and must be progressing
* Prior autologous and/or allogeneic transplant is permitted although transplant must have occurred greater than 90 days prior to registration
* Both men and women of all races and ethnic groups are eligible for this study
* Prior radiation is permitted; however, at least 2 weeks must have elapsed since the completion of prior radiation therapy and patients must have recovered from all radiation-associated toxicities to no greater than grade 1 at the time of registration
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%) is required for eligibility; those patients with lower performance status based solely on bone pain secondary to multiple myeloma are eligible
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelet count >= 75,000 and transfusion independent
* Total bilirubin < 1.5 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x the institutional upper limit of normal
* Ability to understand and the willingness to sign a written informed consent document
* Patients must be able to avoid direct contact with pregnant or nursing women, infants and immunocompromised individuals during the days of Reolysin treatment and for two days after
* Patients must not have known human immunodeficiency virus (HIV) infection or active hepatitis B or C infections
* Systolic cardiac function will be assessed at screening if clinically indicated by history and physical; only patients with left ventricular ejection fraction (LVEF) >= 50% will be eligible for enrollment
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL prior to starting therapy and prior to beginning another cycle (if applicable)
* The effects of Reolysin on the developing human fetus are unknown; for this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) starting 28 days prior to starting the study until at least 90 days following discontinuation of the trial therapy; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patients must agree not to donate blood, sperm/ova during the course of taking protocol therapy and for at least 4 weeks after stopping treatment

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study; patients may be receiving concomitant therapy with bisphosphonates and low dose corticosteroids (e.g., prednisone up to but no more than 10 mg by mouth daily or its equivalent) for symptom management and comorbid conditions; doses of corticosteroid should be stable for at least 7 days prior to study treatment
* Patients who are receiving any other therapeutic investigational agents
* Patients previously treated on clinical trial with Reolysin
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction in the preceding 6 months, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because protocol therapy has the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to protocol treatment of the mother, breastfeeding should be discontinued
* Patients with a "currently active" second malignancy that, in the opinion of the principal investigator, will interfere with patient participation, increase patient risk, shorten survival to < 1 year, or confound data interpretation
* Plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein), and skin changes (POEMS) syndrome
* Concurrent use of complementary or alternative medicines that in the opinion of the principal investigator would confound the interpretation of toxicities and/or antitumor activity of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events | Up to 4 weeks post treatment
  Based on Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Adverse events will be perceived causal relationship to the study therapy.
Maximum tolerated dose of combination carfilzomib and wild-type reovirus | Up to 28 days
  Assessed by CTCAE version 5.0. Maximum tolerated dose defined as the highest dose with fewer than 33% dose limiting toxicities observed in cycle 1 or 2 evaluated using CTCAE version 5.0. Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.
Number of patients who required dose modifications and/or dose delays in subsequent cycles | Up to 4 weeks post treatment
  Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.
Proportion of patients who go off treatment due to adverse reactions of refuse further treatment for lesser toxicities that inhibit their willingness to continue participation on the trial | Up to 4 weeks post treatment
  Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.

SECONDARY OUTCOMES:
Reoviral capsid protein production via immunohistochemical analysis | Up to day 9 of cycle 1
  Will include graphical evaluation of these immunologic correlative markers at baseline as well as at the various timepoints.
Presence and location of intracellular reoviral ribonucleic acid (RNA) assessed by in situ hybridization | Up to day 9 of cycle 1
  Will include graphical evaluation of these immunologic correlative markers at baseline as well as at the various timepoints.
Number and percentage of subjects experiencing objective response | Up to 4 weeks post treatment
  Summary statistics will be computed for baseline biomarkers. The absolute and percent change from baseline will be calculated for each subsequent measurement. Summary statistics will be computed for each collection time point. The objective response rate will be analyzed by using a 95% confidence interval for the proportion responding at trial closure in the treated population.
Clinical benefit endpoint described as that portion of patients experiencing complete response, very good partial response, or partial response | Up to 4 weeks post treatment
  The objective response rate will be analyzed by using a 95% confidence interval for the proportion responding at trial closure in the treated population.
Duration of response | Duration from first observation of partial response to the time of disease progression, up to 4 weeks post treatment
  This time-to-event distribution will be evaluated using the methods of Kaplan and Meier, with a focus on graphical evaluation as well as early timepoint and median estimates of survival distributions.
Progression free survival | Duration from start of treatment to disease progression or death, regardless of cause of death, whichever comes first, up to 2 years
  This time-to-event distribution will be evaluated using the methods of Kaplan and Meier, with a focus on graphical evaluation as well as early timepoint and median estimates of survival distributions.
Time to progression | Time from the start of the treatment until the criteria for disease progression are met, up to 4 weeks post treatment
  This time-to-event distribution will be evaluated using the methods of Kaplan and Meier, with a focus on graphical evaluation as well as early timepoint and median estimates of survival distributions.

OTHER OUTCOMES:
Immunologic correlative markers | Up to 2 years
  Will descriptively summarize the continuous markers quantitatively. Patterns of change in the longitudinal data on these markers will be evaluated in this manner for each of the correlative outcomes of interest. Appropriate transformations of the various correlative markers will be used in the presence of skewed data distributions. Multiple comparison corrections will not be used for these secondary correlative analyses. Peripheral blood will be collected at pretreatment on day 1, day 2, and day 9, 15 and once during days 22-28 of cycle 1, and day 1 of cycle 2 and each successive cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Craig C Hofmeister, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Dona AA, Tandoh T, Nigam L, Singer M, Caserta E, Murtadha M, Zhu Y, Moloudizargari M, Sharma P, Napolitano O, Winchester J, Chowdhury A, Pozhitkov A, Sanchez JF, Vahed H, Marcucci G, Coffey M, Nuovo G, Sborov DW, Pichiorri F, Hofmeister CC. Proteasome inhibition enhances oncolytic reovirus therapy in multiple myeloma independently of its direct cytotoxic effects. J Hematol Oncol. 2025 Jan 20;18(1):1. doi: 10.1186/s13045-024-01645-3. PMID 39828738